CLINICAL TRIAL: NCT00367393
Title: An Open-label Multicenter 12-month Long Term Study on Skin Reconstitution With Pimecrolimus Cream 1% in Adult Patients With Atopic Eczema and Corticosteroid Induced Skin Damage
Brief Title: Reconstitution With Pimecrolimus Cream 1% of Steroid-damaged Skin in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981CDE20
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Atopic Dermatitis
Keywords: Pimecrolimus, skin atrophy, dermoscopy, atopic dermatitis, eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus

ARMS (1):
- 1 (Experimental): Pimecrolimus cream 1%
  Interventions: Drug: Pimecrolimus cream 1%

INTERVENTIONS:
Drug: Pimecrolimus cream 1% — Pimecrolimus cream 1% bid, as needed
  Other Names: ASM981

SUMMARY:
Topical steroid use may lead to skin deterioration and spider veins. This study will examine long-term management of atopic dermatitis (AD) over 12 months with pimecrolimus cream 1% and its effect on skin reconstitution of steroid-damaged skin and disease control.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed AD
* almost clear to mild AD (local IGA [target lesions face and cubital areas] score of 1-3)
* clinically (i.e. to the unaided eye) evident skin atrophy due to long-term topical steroid use
* Dermatophot Score (DPS - composed of skin atrophy and telangiectasia) of 4-6 on at least two target areas

Exclusion Criteria:

* Phototherapy or systemic therapy known or suspected to have an effect on AD within 4 weeks prior to study entry
* Topical therapy known or suspected to have an effect on AD within 7 days prior to study entry or systemic corticosteroids within 4 weeks prior to study entry
* Clinical conditions other than AD that according to investigator can interfere with the Dermatophot evaluation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
• Decrease of the Dermatophot (a combination of a dermatoscope and a camera) score on skin deterioration and spider veins from baseline to end of the study | 48 weeks

SECONDARY OUTCOMES:
• Epidermal thickness by optical coherence tomography at selected investigational centers | 48 weeks
Skin thickness by ultrasound at selected investigational centers | 48 weeks
Epidermal thickness by 3mm punch biopsies (optional) | 48 weeks
Skin metabolism by suction blisters. | 48 weeks
Investigator's Global Assessment (IGA) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharm, Study Chair — Novartis
Locations (1):
- Novartis, Novartis, Germany

REFERENCES:
- [Background] Reference: Thaci D et al TBD. CORTICOSTEROID-INDUCED SKIN DAMAGE IMPROVED WITH PIMECROLIMUS CREAM 1% TREATMENT: A 1-YEAR STUDY IN ADULTS WITH ATOPIC ECZEMA. European Academy of Dermatology and Venereology - 17th Congress. 2008; www.eadv.org